CLINICAL TRIAL: NCT05989113
Title: Evaluation of the Psychometric Qualities of the International Physical Activity Questionnaire-Short Form (IPAQ-SF) in Patients With Lower Limb Amputations (QUAPSY)
Brief Title: Psychometric Qualities IPAQ-SF
Acronym: QUAPSY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FondationbHopale (Other)
Responsible Party: Sponsor
Other Study IDs: HOP23-RIPH3-09
Record Dates: First submitted 2023-04-27; First posted 2023-08-14 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-04

CONDITIONS: Amputation; Lower Extremity Amputation; Gait Analysis; Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower limb amputee patients with devices
  Interventions: Other: Administration of the IPAQ-SF questionnaire

INTERVENTIONS:
Other: Administration of the IPAQ-SF questionnaire — Administration of the IPAQ-SF questionnaire at the patient's consultation and upon return home

SUMMARY:
This is an observational, prospective multicentric study designed to develop medical knowledge.

The aim of the study is to validate the IPAQ-SF questionnaire in a population of lower limb amputee patients.

The questionnaire is administered twice to each patient, once during the consultation and again when they return home. Patients also undergo a 6-minute walk test.

DETAILED DESCRIPTION:
This is an observational, prospective multicentric study designed to develop medical knowledge.

The IPAQ is an internationally validated questionnaire for measuring physical activity in healthy subjects.

The IPAQ-SF (short format of the IPAQ) assesses overall physical activity and sedentary time during the last seven days. The IPAQ-SF has been used in a population of lower limb amputees on several occasions, but no study of its psychometric qualities in application to this population has been performed to date.

The main objective of the study is therefore to gather a set of arguments allowing the IPAQ-SF to be used in the follow-up consultation of patients with lower limb amputations who are fitted with a device.

This would help health professionals to assess the physical activity of this population and to develop physical activity promotion interventions adapted to their needs.

This study is part of the standard management of patients with lower limb amputations and devices. In addition to the clinical data and the result of the 6-minute test from the classical management, the IPAQ-SF questionnaire will be completed twice by the patients included in this study:

* Once during the consultation,
* Once at home.

For the only center equipped (center 01) with inertial sensors, the gait parameters during the 6-minute test will be collected in order to extract fatigue indices.

Upon completion of the IPAQ-SF questionnaire a second time, the patient's participation in the study ends.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a major lower limb amputation: transtibial, transfemoral, hip or knee disarticulation or trans-iliolumbar
* Fitting more than 1 year old
* Age 15-69 years (IPAQ-SF not validated outside these ages)
* All causes of amputation (vascular, traumatic, tumor, infectious...)
* Patient having given their informed consent
* Patient affiliated to a social security system

Exclusion Criteria:

* Subjects with bilateral amputations
* Inability to fully and adequately understand the questionnaire (i.e., cognitive impairment, patient does not speak French)
* Contraindication to the 6-minute walk test (chest pain, palpitations, mental confusion or lack of coordination and balance, dizziness or malaise, intolerable dyspnea, leg cramps or extreme leg muscle fatigue, any other clinically justified reason).
* Patients under legal protection (under guardianship, under curatorship, safeguard of justice)
* Pregnant or breast-feeding woman

Ages: 15 Years to 69 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Lower limb amputee patients with devices
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Correlation of the METs/week questionnaire results with the results of the 6-minute walk test | Data collection during the routine consultation on the day of inclusion
  The results of the IPAQ-SF questionnaire will be expressed in METs/week (Metabolic Equivalent of Task).
  The distance covered by the patient at the end of the 6-minute test will be collected in meters.

SECONDARY OUTCOMES:
Relationships between the patients ability to perform his or her expected daily functions after rehabilitation (MFCL classification, out of 5 points) and the IPAQ-SF score. | Data collection during the routine consultation on the day of inclusion
  The MFCL consists of five ordered categories or 'K-levels' that define increasing functional mobility.
Relationships between the level of amputation and the IPAQ-SF score. | Data collection during the routine consultation on the day of inclusion
  5 levels of amputation :
  * Hip disarticulation
  * Transfemoral amputation
  * Knee disarticulation
  * Transtibial amputation
  * Trans-iliolumbar amputation
Relationships between the patient's weight and the IPAQ-SF score. | Data collection during the routine consultation on the day of inclusion
  Patient's weight in kilogram
Relationships between type of prosthesis and the IPAQ-SF score. | Data collection during the routine consultation on the day of inclusion
Relationships between the age of amputation and the IPAQ-SF score. | Data collection during the routine consultation on the day of inclusion
  Age of amputation in years
Relationships between the physical activity level of lower limb amputee patients and the patient's walking speed measured by inertial units during the 6-minute test. | Data collection during the 6-minute routine consultation test on the day of inclusion
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  Patient's walking speed in meters per second during the 6-minute test.
Relationship between the physical activity level of patients with lower-limb amputations and the patient's average step length measured by inertial units during the 6-minute test. | Data collection during the 6-minute routine consultation test on the day of inclusion
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  Patient's average step length in centimeters during the 6-minute test.
Relationship between the physical activity level of patients with lower-limb amputations and the average width of the patient's step measured by inertial units during the 6-minute test. | Data collection during the 6-minute routine consultation test on the day of inclusion
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  Patient's average step width in centimeters during the 6-minute test.
Relationship between the physical activity level of patients with lower-limb amputations and the patient's walking cadence measured by inertial units during the 6-minute test. | Data collection during the 6-minute routine consultation test on the day of inclusion
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  Number of steps per minute during the 6-minute test.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Charlaté, Principal Investigator — Fondation Hopale
Locations (3):
- France (3):
  - Institut Calvé, Berck
  - CHRU Lille - Hôpital Swynghedauw, Lille
  - CRF les HAUTOIS- CRO, Oignies

REFERENCES:
- See also: Deans S, Burns D, McGarry A, et al. Motivations and barriers to prosthesis users participation in physical activity, exercise and sport: a review of the literature. Prosthet Orthot Int. 2012;36:260-269. — https://doi.org/10.1177/0309364612437905
- See also: Wetterhahn, K. A., Hanson, C., & Levy, C. E. (2002). Effect of participation in physical activity on body image of amputees. American journal of physical medicine & rehabilitation, 81(3), 194-201. — https://doi.org/10.1097/00002060-200203000-00007
- See also: Melo, V. H., Sousa, R. A. L., Improta-Caria, A. C., & Nunes, M. A. P. (2021). Physical activity and quality of life in adults and elderly individuals with lower limb amputation. Revista da Associacao Medica Brasileira (1992), 67(7), 985-990 — https://doi.org/10.1590/1806-9282.20210382
- See also: da Silva, R., Rizzo, J. G., Gutierres Filho, P. J., Ramos, V., & Deans, S. (2011). Physical activity and quality of life of amputees in southern Brazil. Prosthetics and orthotics international, 35(4), 432-438. — https://doi.org/10.1177/0309364611425093
- See also: Shema-Shiratzky (2019). Deterioration of specific aspects of gait during the instrumented 6-min walk test among people with multiple sclerosis. Jou — https://doi.org/10.1007/s00415-019-09500-z
- See also: Van Schooten (2016). Daily-Life Gait Quality as Predictor of Falls in Older People: A 1-Year Prospective Cohort Study. — https://doi.org/10.1371/journal.pone.0158623